CLINICAL TRIAL: NCT04708145
Title: Long-Term Efficacy and Safety of Intravitreal Aflibercept Injections for the Treatment of Diabetic Retinopathy for Subjects Who Completed the 2-Year PANORAMA Trial
Acronym: VOYAGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Greater Houston Retina Research (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Clinical Trials Resource Group, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VOYAGE
Record Dates: First submitted 2021-01-06; First posted 2021-01-13 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Study eyes without PRP from the PANORAMA trial. Subjects will be evaluated every 16 weeks and treated if DRSS level is 47 or worse as determined by the treating investigator.
  Subjects may be evaluated every 8 weeks if a 2-step DRSS level worsening compared to the last protocol-scheduled 16-week visit occurs, the DRSS level is 53 or worse, or if a subject has active PDR. Visits can continue every 8 weeks until there is no active PDR, and the DRSS improves to the level observed at the visit before the subject began being seen at 8-week intervals. Thereafter, visits will continue at 16 week intervals.
  Interventions: Drug: Aflibercept Injection
- Group 2 (Experimental): Study eyes with PRP from the PANORAMA trial. Subjects will be evaluated every 16 weeks and treated if the neovascular disease process is active and stable (not new or worse) as determined by the treating investigator. If the neovascular disease is inactive, no treatment will be given.
  If new or worsening neovascularization develops, subjects may be seen and treated every 8 weeks until the neovascular disease is stable or inactive, at which time the interval between visits will increase to 16 weeks.
  Interventions: Drug: Aflibercept Injection

INTERVENTIONS:
Drug: Aflibercept Injection — Intravitreal 2mg aflibercept injection
  Other Names: Eylea

SUMMARY:
The VOYAGE trial will assess diabetic retinopathy severity scale (DRSS) levels, through 112 weeks, while being managed with aflibercept as needed, among subjects who completed the 2-year PANORAMA trial (VGFTe-OD-1411) and were treated in a clinical setting prior to joining the VOYAGE study.

DETAILED DESCRIPTION:
This phase 4 study is designed to assess the need for ongoing 2 mg intravitreal aflibercept injections (IAI) for subjects who completed the 2-year PANORAMA (VGFTe-OD-1411) trial for the management of diabetic retinopathy (DR). Sites will be considered for VOYAGE if they have 4 or more subjects from PANORAMA able to participate.

Relevant data from all participating subjects will be collected and reported retrospectively for the period between PANORAMA study exit and VOYAGE study enrollment.

For the prospective portion of the study, eyes will be assigned to 1 of 2 groups, eyes without panretinal photocoagulation (PRP) and eyes with PRP.

Group 1: Subjects with study eyes without PRP will be seen every 16 weeks (Q16W) and treated with IAI on a flexible treatment regimen based on their DRSS level. An injection will be given at each 16-week visit when the DRSS level is 47 or worse. If the DRSS level is better than 47, for example level 43 or 35, the study eye will not be treated. DRSS level will be determined by the investigator, based on ophthalmic exam and fundus photography (FP) compared to prior imaging when available.

Every 8 week visits can be performed under specific circumstances:

* If a subject has a 2-step DRSS level worsening compared to the last protocol-scheduled 16-week visit (for example the week-16 or week-32 visit) and/or the DRSS level is 53 or worse OR
* If a subject has active proliferative DR (PDR)

Under both of these circumstances, IAI will be administered as scheduled and the subject can be seen and treated every 8 weeks (Q8W) with IAI. Under both of these circumstances, Q8W visits and Q8W IAI treatments can be continued until there is no active PDR and the DRSS improves to the level observed at the visit before the subject began being seen at 8-week intervals.

Group 2: Subjects with study eyes with PRP will be seen Q16W and treated with IAI on a flexible treatment regimen based on activity of the neovascular disease process as assessed by the treating investigator based on ophthalmic exam and/or FP compared to prior imaging when available. If the neovascular disease is inactive, no treatment will be given. If the neovascular disease is active and stable (not new or worse), the subject will be treated with intravitreal (IVT) IAI at the Q16W interval. If new or worsening neovascular disease develops, subjects may be seen and treated Q8W until the neovascular disease is stable or inactive at which time the interval between visits will increase to 16 weeks.

Subjects in both groups will be evaluated for efficacy, using best corrected visual acuity (BCVA) using the 4-meter ETDRS protocol with normal-luminance, Humphrey Visual Field (HVF), National Eye Institute (NEI) Visual Function Questionnaire (VFQ) 25, spectral domain optical coherence tomography (SD-OCT), optical coherence tomography angiography (OCT-A), FP, and fluorescein angiography (FA), and for ocular and systemic safety (including ophthalmic exams and laboratory assessments) through week 112.

Subjects who develop new or worsening PDR, including anterior segment neovascularization (ASNV), or center-involved DME may qualify for rescue treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled and completed PANORAMA (VGFTe-OD-1411) clinical trial
2. Willing and able to comply with clinic visits and study-related procedures
3. Provide signed informed consent

Exclusion Criteria:

1. Any prior systemic anti-vascular endothelial growth factor (VEGF) treatment or IVT anti-VEGF treatment in the study eye within 21 days of baseline
2. Any intra- or periocular corticosteroid treatment in the study eye within 3 months of baseline
3. Any intraocular sustained-release treatment, implantable device, or gene therapy in the study eye
4. Pregnant or breastfeeding women
5. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening/baseline; intrauterine device (IUD); bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly).

   * Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrhoeic for at least 12 months in order not to be considered of childbearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
DRSS Level Achievement in the VOYAGE study | 112 weeks
  Proportion of subjects achieving a DRSS level of 43 or less in the VOYAGE study.

SECONDARY OUTCOMES:
DRSS Level Achievement in the PANORAMA study | 112 weeks
  Proportion of subjects achieving a DRSS level of 43 or less from the completion of the PANORAMA study
DRSS Level Improvement | 112 weeks
  Proportion of subjects with stable, worsened, or improved DRSS level from baseline to week 48 and baseline to week 112 compared to the DRSS at the baseline of the VOYAGE trial and the DRSS at the last visit of the PANORAMA trial.
Injection Frequency | 112 weeks
  Mean and median number of IVT aflibercept injections (with and without IAI given for DME)
Subjects without Treatment | 112 weeks
  Proportion of subjects receiving 0 injections
PDR Events | 112 weeks
  Percentage of subjects over time who develop a new PDR event
Center-Involved Diabetic Macular Edema Development | 112 weeks
  Percentage of subjects over time who develop center-involved (CI) DME
Change in Visual Acuity | 112 weeks
  Mean change in ETDRS BCVA from baseline
Change in Central Retinal Thickness | 112 weeks
  Mean change in central retinal thickness from baseline
Change in Area of Nonperfusion | 112 weeks
  Change in total area of retinal capillary non-perfusion from baseline
Changes in Visual Function (HVF) | 112 weeks
  Changes in visual function outcomes from Humphrey Visual Field from baseline
Changes in Visual Function | 112 weeks
  Changes in visual function outcomes NEI VFQ-25 from baseline
Incidence of Adverse Events | 112 weeks
  Incidence and severity of ocular and systemic adverse events from baseline

CONTACTS AND LOCATIONS:
Locations (14):
- United States (13):
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Central Florida Retina Center, Orlando, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Marietta Eye Clinic, Marietta, Georgia
  - John Kenyon American Eye Institute, New Albany, Indiana
  - Cumberland Valley Retina Consultants, P.C., Hagerstown, Maryland
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Palmetto Retina Center, LLC - Florence, Florence, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Charles Retina Institute, Germantown, Tennessee
  - Retina Consultants of Texas, Bellaire, Texas
  - Valley Retina Institute, Harlingen, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
- Emanuelli Research and Development Center, LLC, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kempen JH, O'Colmain BJ, Leske MC, Haffner SM, Klein R, Moss SE, Taylor HR, Hamman RF; Eye Diseases Prevalence Research Group. The prevalence of diabetic retinopathy among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):552-63. doi: 10.1001/archopht.122.4.552. PMID 15078674
- [Background] Leasher JL, Bourne RR, Flaxman SR, Jonas JB, Keeffe J, Naidoo K, Pesudovs K, Price H, White RA, Wong TY, Resnikoff S, Taylor HR; Vision Loss Expert Group of the Global Burden of Disease Study. Global Estimates on the Number of People Blind or Visually Impaired by Diabetic Retinopathy: A Meta-analysis From 1990 to 2010. Diabetes Care. 2016 Sep;39(9):1643-9. doi: 10.2337/dc15-2171. PMID 27555623
- [Background] Bourne RR, Stevens GA, White RA, Smith JL, Flaxman SR, Price H, Jonas JB, Keeffe J, Leasher J, Naidoo K, Pesudovs K, Resnikoff S, Taylor HR; Vision Loss Expert Group. Causes of vision loss worldwide, 1990-2010: a systematic analysis. Lancet Glob Health. 2013 Dec;1(6):e339-49. doi: 10.1016/S2214-109X(13)70113-X. Epub 2013 Nov 11. PMID 25104599
- [Background] Fong DS, Girach A, Boney A. Visual side effects of successful scatter laser photocoagulation surgery for proliferative diabetic retinopathy: a literature review. Retina. 2007 Sep;27(7):816-24. doi: 10.1097/IAE.0b013e318042d32c. PMID 17891003
- [Background] Ferris F. Early photocoagulation in patients with either type I or type II diabetes. Trans Am Ophthalmol Soc. 1996;94:505-37. PMID 8981711
- [Background] Diabetic Retinopathy Clinical Research Network; Elman MJ, Aiello LP, Beck RW, Bressler NM, Bressler SB, Edwards AR, Ferris FL 3rd, Friedman SM, Glassman AR, Miller KM, Scott IU, Stockdale CR, Sun JK. Randomized trial evaluating ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2010 Jun;117(6):1064-1077.e35. doi: 10.1016/j.ophtha.2010.02.031. Epub 2010 Apr 28. PMID 20427088
- [Background] Nguyen QD, Brown DM, Marcus DM, Boyer DS, Patel S, Feiner L, Gibson A, Sy J, Rundle AC, Hopkins JJ, Rubio RG, Ehrlich JS; RISE and RIDE Research Group. Ranibizumab for diabetic macular edema: results from 2 phase III randomized trials: RISE and RIDE. Ophthalmology. 2012 Apr;119(4):789-801. doi: 10.1016/j.ophtha.2011.12.039. Epub 2012 Feb 11. PMID 22330964
- [Background] Korobelnik JF, Do DV, Schmidt-Erfurth U, Boyer DS, Holz FG, Heier JS, Midena E, Kaiser PK, Terasaki H, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Brown DM. Intravitreal aflibercept for diabetic macular edema. Ophthalmology. 2014 Nov;121(11):2247-54. doi: 10.1016/j.ophtha.2014.05.006. Epub 2014 Jul 8. PMID 25012934
- [Background] Writing Committee for the Diabetic Retinopathy Clinical Research Network; Gross JG, Glassman AR, Jampol LM, Inusah S, Aiello LP, Antoszyk AN, Baker CW, Berger BB, Bressler NM, Browning D, Elman MJ, Ferris FL 3rd, Friedman SM, Marcus DM, Melia M, Stockdale CR, Sun JK, Beck RW. Panretinal Photocoagulation vs Intravitreous Ranibizumab for Proliferative Diabetic Retinopathy: A Randomized Clinical Trial. JAMA. 2015 Nov 24;314(20):2137-2146. doi: 10.1001/jama.2015.15217. PMID 26565927
- [Background] Diabetic Retinopathy Clinical Research Network; Wells JA, Glassman AR, Ayala AR, Jampol LM, Aiello LP, Antoszyk AN, Arnold-Bush B, Baker CW, Bressler NM, Browning DJ, Elman MJ, Ferris FL, Friedman SM, Melia M, Pieramici DJ, Sun JK, Beck RW. Aflibercept, bevacizumab, or ranibizumab for diabetic macular edema. N Engl J Med. 2015 Mar 26;372(13):1193-203. doi: 10.1056/NEJMoa1414264. Epub 2015 Feb 18. PMID 25692915
- [Background] Sivaprasad S, Prevost AT, Vasconcelos JC, Riddell A, Murphy C, Kelly J, Bainbridge J, Tudor-Edwards R, Hopkins D, Hykin P; CLARITY Study Group. Clinical efficacy of intravitreal aflibercept versus panretinal photocoagulation for best corrected visual acuity in patients with proliferative diabetic retinopathy at 52 weeks (CLARITY): a multicentre, single-blinded, randomised, controlled, phase 2b, non-inferiority trial. Lancet. 2017 Jun 3;389(10085):2193-2203. doi: 10.1016/S0140-6736(17)31193-5. Epub 2017 May 7. PMID 28494920
- [Background] Mazhar K, Varma R, Choudhury F, McKean-Cowdin R, Shtir CJ, Azen SP; Los Angeles Latino Eye Study Group. Severity of diabetic retinopathy and health-related quality of life: the Los Angeles Latino Eye Study. Ophthalmology. 2011 Apr;118(4):649-55. doi: 10.1016/j.ophtha.2010.08.003. Epub 2010 Oct 29. PMID 21035872
- [Background] Klein R, Knudtson MD, Lee KE, Gangnon R, Klein BE. The Wisconsin Epidemiologic Study of Diabetic Retinopathy XXIII: the twenty-five-year incidence of macular edema in persons with type 1 diabetes. Ophthalmology. 2009 Mar;116(3):497-503. doi: 10.1016/j.ophtha.2008.10.016. Epub 2009 Jan 22. PMID 19167079
- [Background] Fundus photographic risk factors for progression of diabetic retinopathy. ETDRS report number 12. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):823-33. PMID 2062515
- [Background] Klein R, Klein BE, Moss SE. How many steps of progression of diabetic retinopathy are meaningful? The Wisconsin epidemiologic study of diabetic retinopathy. Arch Ophthalmol. 2001 Apr;119(4):547-53. doi: 10.1001/archopht.119.4.547. PMID 11296020
- [Background] Wilkinson CP, Ferris FL 3rd, Klein RE, Lee PP, Agardh CD, Davis M, Dills D, Kampik A, Pararajasegaram R, Verdaguer JT; Global Diabetic Retinopathy Project Group. Proposed international clinical diabetic retinopathy and diabetic macular edema disease severity scales. Ophthalmology. 2003 Sep;110(9):1677-82. doi: 10.1016/S0161-6420(03)00475-5. PMID 13129861
- [Background] Brown DM, Schmidt-Erfurth U, Do DV, Holz FG, Boyer DS, Midena E, Heier JS, Terasaki H, Kaiser PK, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Korobelnik JF. Intravitreal Aflibercept for Diabetic Macular Edema: 100-Week Results From the VISTA and VIVID Studies. Ophthalmology. 2015 Oct;122(10):2044-52. doi: 10.1016/j.ophtha.2015.06.017. Epub 2015 Jul 18. PMID 26198808
- [Background] Brown DM, Nguyen QD, Marcus DM, Boyer DS, Patel S, Feiner L, Schlottmann PG, Rundle AC, Zhang J, Rubio RG, Adamis AP, Ehrlich JS, Hopkins JJ; RIDE and RISE Research Group. Long-term outcomes of ranibizumab therapy for diabetic macular edema: the 36-month results from two phase III trials: RISE and RIDE. Ophthalmology. 2013 Oct;120(10):2013-22. doi: 10.1016/j.ophtha.2013.02.034. Epub 2013 May 22. PMID 23706949
- [Background] Ip MS, Domalpally A, Hopkins JJ, Wong P, Ehrlich JS. Long-term effects of ranibizumab on diabetic retinopathy severity and progression. Arch Ophthalmol. 2012 Sep;130(9):1145-52. doi: 10.1001/archophthalmol.2012.1043. PMID 22965590
- [Background] Ip MS, Domalpally A, Sun JK, Ehrlich JS. Long-term effects of therapy with ranibizumab on diabetic retinopathy severity and baseline risk factors for worsening retinopathy. Ophthalmology. 2015 Feb;122(2):367-74. doi: 10.1016/j.ophtha.2014.08.048. Epub 2014 Nov 18. PMID 25439595
- [Background] Bressler SB, Liu D, Glassman AR, Blodi BA, Castellarin AA, Jampol LM, Kaufman PL, Melia M, Singh H, Wells JA; Diabetic Retinopathy Clinical Research Network. Change in Diabetic Retinopathy Through 2 Years: Secondary Analysis of a Randomized Clinical Trial Comparing Aflibercept, Bevacizumab, and Ranibizumab. JAMA Ophthalmol. 2017 Jun 1;135(6):558-568. doi: 10.1001/jamaophthalmol.2017.0821. PMID 28448655
- [Background] Wykoff CC, Le RT, Khurana RN, Brown DM, Ou WC, Wang R, Clark WL, Boyer DS; ENDURANCE Study Group. Outcomes With As-Needed Aflibercept and Macular Laser Following the Phase III VISTA DME Trial: ENDURANCE 12-Month Extension Study. Am J Ophthalmol. 2017 Jan;173:56-63. doi: 10.1016/j.ajo.2016.09.029. Epub 2016 Oct 1. PMID 27702624
- [Derived] Zhou AW, Teagle GM, Baumann LM, Cao JA, Emanuelli A, Hu AY, Berger AS, Major JC Jr, Lee SY, Huddleston SM, Gonzalez VH, Clark WL, Liao DS, Kingsley RM, Lazarus HS, Payne JF, Feinstein EG, Meleth AD, Patel SB, Fan KC, Berliner AJ, Moini H, Niu X, Ip MS, Sadda SR, Al-Khersan H, Wykoff CC. Intravitreal Aflibercept for the Treatment of Diabetic Retinopathy Among Patients Who Completed PANORAMA: 1-Year Outcomes from the VOYAGE Extension Study. J Pers Med. 2025 Nov 14;15(11):555. doi: 10.3390/jpm15110555. PMID 41295257
- See also: World Health Organization (WHO). Global Report on Diabetes. 2016. — http://apps.who.int/iris/bitstream/10665/204871/1/9789241565257_eng.pdf?ua=1&ua=1
- See also: Study of the Efficacy and Safety of Intravitreal (IVT) Aflibercept for the Improvement of Moderately Severe to Severe Nonproliferative Diabetic Retinopathy (NPDR) (PANORAMA) — https://www.clinicaltrials.gov/ct2/show/NCT02718326?term=PANORAMA&rank=5